CLINICAL TRIAL: NCT02381366
Title: A Phase I/II, Open-Label Dose Escalation Trial to Evaluate the Safety and Efficacy of Two Dose Levels of PNEUMOSTEM® in Premature Infants at High Risk for Bronchopulmonary Dysplasia (BPD)
Brief Title: Safety and Efficacy of PNEUMOSTEM® in Premature Infants at High Risk for Bronchopulmonary Dysplasia (BPD) - a US Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medipost, Inc. (Industry)
Collaborators: Medipost Co Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MD-BPD-US001
Record Dates: First submitted 2015-02-15; First posted 2015-03-06 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Mesenchymal Stem Cells; Human Umbilical Cord Blood; Premature Infants; Bronchopulmonary Dysplasia; Chronic Lung Disease; Cell Therapy
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PNEUMOSTEM® (Experimental): Dose A: PNEUMOSTEM® 10 million cells per kg Dose B: PNEUMOSTEM® 20 million cells per kg
  Interventions: Biological: Human Umbilical Cord Blood Derived-Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Human Umbilical Cord Blood Derived-Mesenchymal Stem Cells — Human Umbilical Cord Blood Derived-Mesenchymal Stem Cells:
  Dose A: 10 million cells per kg / Dose B: 20 million cells per kg
  Other Names: PNEUMOSTEM®

SUMMARY:
PNEUMOSTEM® consists of ex vivo cultured allogeneic, unrelated, human umbilical cord blood-derived mesenchymal stem cells (hUCB-MSCs) and it is intended for use as a cellular therapy product for prevention of Bronchopulmonary Dysplasia (BPD). This study is an open-label, single-center, dose escalation study to evaluate of safety and efficacy of PNEUMOSTEM® in premature infants at high risk for BPD.

ELIGIBILITY:
Inclusion Criteria:

* A male or female infant whose postnatal age is 3 to 14 days, inclusive (for treatment between 5 and 14 days after birth)
* A subject whose gestational age is between 23 and 28 weeks (23 weeks ≤ gestational age (GA) < 28 weeks)
* A subject whose birth weight is between 500g and 1000g, inclusive
* A subject who is intubated and receiving mechanical ventilation within 5-14 days after birth, with a fraction of inspired oxygen (FiO2) of 0.25 or greater at Screening
* A subject who has had either a deterioration or no change in the setting of mechanical ventilation within the 24 hours before trial enrollment
* A subject whose parent/guardian can give a written informed consent

Exclusion Criteria:

* A subject who has a congenital heart defect, except for patent ductus arteriosus (PDA), atrial septal defect (ASD) or a small, restrictive ventricular septal defect (VSD)
* A subject who has a serious malformation of the lung such as pulmonary hypoplasia/aplasia congenital diaphragmatic hernia, or other congenital lung anomaly
* A subject who has a chromosomal abnormality (e.g., Trisomy 18, Trisomy 13 or Trisomy 21) or a severe congenital malformation (e.g., hydrocephalus and encephalocele, tracheo-esophageal fistula, abdominal wall defects, and major renal anomalies)
* A subject who has had a severe congenital infectious disease (i.e., herpes, toxoplasmosis rubella, syphilis, HIV, etc.)
* A subject who has evidence of severe sepsis or septic shock due to an active infection at Screening
* A subject who underwent a surgical procedure within 72 hours before study drug administration or who is anticipated to have a surgical procedure within 72 hours before or following study drug administration
* A subject who was administered surfactant within 24 hours before study drug administration
* A subject who has had a bilateral grade 3 or 4 intracranial hemorrhage
* A subject who has active pulmonary hemorrhage or an active air leak syndrome at Screening
* A subject who is currently participating in any other interventional clinical trial
* A subject who is, in the opinion of the Principal Investigator, considered inappropriate for the trial due to any reasons other than those listed above

Ages: 3 Days to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse reactions for 84 days after treatment | 84 days

SECONDARY OUTCOMES:
Number of participants with adverse reactions between 84 days after treatment and 20 months of corrected age | Between 84 days after treatment and 20 months of corrected age
Incidence of moderate/severe BPD or death at 36 weeks postmenstrual age (PMA) | 36 weeks PMA
Hospital Re-admission between 84 days after treatment until 20 months of corrected age | Between 84 days after treatment and 20 months of corrected age
Bayley Scales of Infant and Toddler Development between 84 days after treatment until 20 months of corrected age | Between 84 days after treatment and 20 months of corrected age

CONTACTS AND LOCATIONS:
Overall Officials: Steven Powell, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Powell SB, Silvestri JM. Safety of Intratracheal Administration of Human Umbilical Cord Blood Derived Mesenchymal Stromal Cells in Extremely Low Birth Weight Preterm Infants. J Pediatr. 2019 Jul;210:209-213.e2. doi: 10.1016/j.jpeds.2019.02.029. Epub 2019 Apr 13. PMID 30992220